CLINICAL TRIAL: NCT04693585
Title: Development and Pilot Test of an mHealth Interactive Education and Social Support Intervention for Improving Postnatal Health - Phase 2
Brief Title: Development and Pilot Test of a Postnatal mHealth Intervention - Phase 2
Acronym: MESSAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Indraprastha Institute of Information Technology Delhi (Other); Survival for Women and Children Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R21HD101786-A; R21HD101786 (NIH)
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Health Attitude; Knowledge, Attitudes, Practice; Post Partum Depression; Acceptability of Health Care
MeSH Terms: conditions — Behavior; Depression, Postpartum; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: The three intervention modalities to be tested include: real-time live voice calls versus audio/video recording; text-based, asynchronous, on-demand social support; and standard of postnatal care (3 visits in first 7 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: live support (Experimental): Real-time live voice call plus standard of postnatal care.
  Interventions: Behavioral: MESSSSAGE - live
- Arm 2: asynchronous support (Experimental): Text-based, asynchronous, on-demand social support plus standard of postnatal care
  Interventions: Behavioral: MESSSSAGE - asynchronous
- Arm 3: both live and asynchronous support (Experimental): Real-time live voice call plus standard of postnatal care; text-based, asynchronous, on-demand social support plus standard of postnatal care
  Interventions: Behavioral: MESSSSAGE - live; Behavioral: MESSSSAGE - asynchronous
- Arm 4: control (No Intervention): Standard of postnatal care.

INTERVENTIONS:
Behavioral: MESSSSAGE - live — mHealth education and social support intervention, synchronous via call
  Arms: Arm 1: live support; Arm 3: both live and asynchronous support
Behavioral: MESSSSAGE - asynchronous — mHealth education and social support intervention, asynchronous via text
  Arms: Arm 2: asynchronous support; Arm 3: both live and asynchronous support

SUMMARY:
The goal of the study is to assess the feasibility and acceptability of the optimized MeSSSSage intervention which was developed and revised based on the results of our initial pilot testing. The investigators will conduct a controlled 4-arm factorial design randomized study to test the feasibility, acceptability and preliminary effectiveness of several intervention modalities over a 6-month period.

DETAILED DESCRIPTION:
Most mHealth interventions for maternal and child health (MCH) in low and middle-income countries, including India, have focused on unidirectional and non-interactive approaches, primarily text messaging. However, ample evidence suggests that provider-led, interactive educational programming and social support are key for improving health behaviors and outcomes. Thus innovative mHealth approaches that promote interactive education and facilitate social support have great potential to improve MCH outcomes. The two-phase development of MeSSSSage include sPhase 1: exploratory development on functions and platforms and Phase 2: a mixed-methods randomized pilot study using a factorial design of specific intervention functions and platforms confirmed in Phase 1. Study activities described herein are associated with Phase 1. The study's specific aim is: To test the optimized intervention to understand the feasibility, acceptability and preliminary effectiveness of several intervention modalities among postnatal women in rural India. In Phase 2, the investigators conduct a randomized factorial design to understand the contribution to various intervention modalities on feasibility, accessibility and preliminary effectiveness. Data are collected via quantitative participant survey (baseline and endline) including sociodemographic characteristics and knowledge about maternal and infant health, self-efficacy, and perceived social norms regarding MCH-related health promoting behaviors (baseline) acceptability questions such as women's satisfaction with and perceptions of MeSSSSage, maternal and infant knowledge-, behavior-, and health-related questions including about breastfeeding, complementary food introduction, immunization, family planning uptake, maternal physical and mental health, etc. The investigators will validate self-report with health records. The investigators will conduct in-depth interviews among a purposive sample of 30 women to understand: mobile technology familiarity prior to intervention, perspectives on intervention and challenges, structure of intervention (group, individual), content, perspectives on the text-based component, relationship with other participants, perspective on the moderator, postnatal period health related concerns, sources of support (social and informational), recommendations. Other assessment will include technological data from, and group moderator surveys and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal (within 2 weeks)
* 18+ years old

Exclusion Criteria:

* Women below 18 years of age
* Women with high risk pregnancies
* Women who delivered preterm, suffer severe maternal complications or they or their baby are otherwise sick in the first week

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison M El Ayadi, ScD, Principal Investigator — University of California, San Francisco; Nadia G Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Post Graduate Institute for Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox V, Sharma P, Verma GS, Gill N, Diamond-Smith NG, Duggal M, Kumar V, Bagga R, Kaur J, Singh P, El Ayadi AM. User acceptability and perceived impact of a mobile interactive education and support group intervention to improve postnatal health care in northern India: a qualitative study. BMC Med Inform Decis Mak. 2025 Feb 20;25(1):93. doi: 10.1186/s12911-025-02935-7. PMID 39980038

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Synchronous and Asynchronous Support: Synchronous: Real-time live voice or video call Asynchronous: Audio-based education via mobile application or interactive voice response on-demand Other: standard of postnatal care
- Arm 2: Asynchronous Support: Asynchronous: Audio-based education via mobile application or interactive voice response on-demand Other: standard of postnatal care
- Arm 3: Control: Other: Standard of postnatal care.
Period: Overall Study
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Started | 120 | 40 | 41
Completed | 94 | 28 | 13
Not Completed | 26 | 12 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control | Total
Number analyzed (Participants) | 120 | 40 | 41 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (3.7) | 26.1 (3.4) | 26.8 (4.9) | 26.6 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 40 | 41 | 201
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 120 | 40 | 41 | 201
Region of Enrollment [Number; unit: participants]
  India | 120 | 40 | 41 | 201

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Being Satisfied or Very Satisfied About Their Overall Intervention Experience
Description: Number of participants reporting being "satisfied" or "very satisfied" with their overall intervention experience, assessed through a five-point Likert scale at six months.
Time Frame: 6 months
Population: Control group participants did not answer questions about intervention experience
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 94 | 28 | 0
Participants | 90 | 19 |

2. Primary Outcome: Number of Participants Engaging in Group Call Intervention
Description: Number of participants who engaged in weekly group call intervention activities by 6 months
Time Frame: 6 months
Population: Group call intervention activities only relevant to arm 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 120 | 0 | 0
Participants | 37 |  |

3. Secondary Outcome: Number of Participants With Knowledge on Maternal and Neonatal Danger Signs, Best Practices for Infant Care, Family Planning.
Description: Number of participants correctly identifying at least 80% of knowledge on maternal and neonatal danger signs, best practices for infant care, and family planning at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 94 | 28 | 13
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Exclusively Breastfeeding
Description: Number of participants who exclusively breastfed their infants through 6 months of age
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 94 | 28 | 13
Participants | 79 | 18 | 11

5. Secondary Outcome: Number of Participants Reporting Postpartum Depression
Description: Number of participants reporting postpartum depression symptoms at six months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 94 | 28 | 13
Participants | 43 | 10 | 5

6. Secondary Outcome: Number of Participants Who Adopted Postpartum Family Planning
Description: Number of participants who started a modern contraceptive methods within 6 months postpartum
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
Number analyzed (Participants) | 94 | 28 | 13
Participants | 67 | 14 | 10

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Arm 1: Synchronous and Asynchronous Support | Arm 2: Asynchronous Support | Arm 3: Control
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/28 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/28 | 0/13
Other Adverse Events (participants affected / at risk) | 0/94 | 0/28 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04693585/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04693585/SAP_001.pdf